CLINICAL TRIAL: NCT03040245
Title: Measuring the Impact of the French Version of the Whiplash Book on Both Treatment Approach and Fears and Beliefs Among Emergency Physicians
Brief Title: Measuring the Impact of the French Version of the Whiplash Book
Acronym: WHIPLASH
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CH Aurillac (Unknown); Jacques Lacarin Hospital Center (Other); CH Moulins (Unknown); CH Montluçon (Unknown); CH Issoire (Unknown); CH Thiers (Unknown); CH Ambert (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU 298
Record Dates: First submitted 2017-01-13; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Whiplash Trauma
Keywords: Emergency physician; Whiplash Book; Whiplash trauma; Fears; Beliefs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (2):
- intervention group: The intervention group was instructed to complete the questionnaires at least 48 hours after the intervention that is, after reading the information booklet
  Interventions: Behavioral: Whiplash book
- control group: The same items were included as in the initial folder, with an additional questionnaire enabling the intervention group to qualitatively assess the information booklet. If there was no response, reminders were sent by email, then by telephone, and lastly by post.
  Interventions: Behavioral: Whiplash book

INTERVENTIONS:
Behavioral: Whiplash book

SUMMARY:
Whiplash trauma and the resulting whiplash associated disorders have been the subject of much attention in the scientific literature and remain a major public health problem.

The most commonly encountered symptoms are neck pain, headache, low back pain, shoulder pain, as well as visual impairment. It is not unusual for neck pain to become chronic, and when this occurs, there may be serious consequences on a social, professional and financial level.

Even though the role of the initial episode should not be ignored, progression to chronic pain is probably multifactorial and, like non-specific low back pain, psycho-social factors, and in particular patient fears and belief, seem to play a relevant role, as do environmental factors. The professional consensus is that it is useful to provide targeted information at an early stage in whiplash settings in order to reduce mistaken fears and beliefs. A preliminary study enabled the investigators to validate a French version of an information booklet that draws on validated data from evidence-based medicine. The booklet was "Le guide du coup de fouet cervical," the French version of The Whiplash Book. This study showed that fears and beliefs were considerably high in a population without neck problems who were working in hospitals. It also revealed that simply providing information could help lessen them.

Management following whiplash injury can make use of the recommendations as published in the literature. Healthcare professionals must reassure and educate their patients that post-traumatic pain is normal, and that they need to remain active and maintain physical activity in order to improve their prognosis.

Only very few studies have evaluated the adherence of physicians or healthcare professionals to the guidelines and to ways of changing their approach to treatment.

The main aim of this study was to determine what fears and beliefs physicians have about the consequences of whiplash. The secondary aim was to measure the impact of a validated information booklet on emergency physicians' approach to management following a whiplash injury.

DETAILED DESCRIPTION:
Once each of the department heads and the different physicians concerned had given their agreement to take part in the study, an initial questionnaire folder (containing the WBQ and FABQ) was sent by email and by post to each of the physicians drawn by randomization. Upon inclusion, demographic data was collected from the physicians (gender, age, place of practice, and length of time in practice), as well as any personal or family history of neck pain or whiplash. The physicians were also asked how often they encountered cases of whiplash.

Information about knowledge of whiplash injury was also sought. This included continuing medical training or recent reading (within the previous 3 years), and in particular knowledge of the different severity grades established by the Quebec Task Force classification, the radiologic recommendations of the Canadian C-Spine Rule, and lastly the latest HAS recommendation on physical therapy in post-whiplash neck pain.

Once the first questionnaire folder had been completed, a second folder was then sent to all physicians participating in the study. The intervention group was instructed to complete the questionnaires at least 48 hours after the intervention that is, after reading the information booklet.

The same items were included as in the initial folder, with an additional questionnaire enabling the intervention group to qualitatively assess the information booklet. If there was no response, reminders were sent by email, then by telephone, and lastly by post.

ELIGIBILITY:
Inclusion Criteria:

* - Both sexes
* Emergency medicine doctors
* Doctors has given its consent to participate in the study

Exclusion Criteria:

* no criteria

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: emergency physicians
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
assessment of fears and beliefs in the sample of physicians tested using questionnaire WBQ (whiplash belief questionnaire) | 48 hours after reading the information booklet
  For each statement, the physician must express his or her level of agreement or disagreement, with a score that varies from 9 to 45. The higher the score, the stronger the beliefs
assessment of fears and beliefs in the sample of physicians tested using the FABQ (Fear Avoidance Belief questionnaire) | 48 hours after reading the information booklet
  The FABQ (Fear Avoidance Belief questionnaire) comprises two independent scales: the physical activity FABQ and work FABQ

SECONDARY OUTCOMES:
Measurement of the impact of a validated information booklet on emergency physicians' approach to management following a whiplash injury. | 10 days for control group or minimum 48 hours after reading the information booklet for interventional group
Non-pharmacological management of a whiplash injury | 10 days for control group or minimum 48 hours after reading the information booklet for interventional group
  Non-pharmacological management of a whiplash injury estimated by :
  * Prescription of necklace (yes/no (%)) If yes, duration of prescription
  * Prescription of physiotherapy sessions (%)
  * Work cessation yes/no (%)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France